CLINICAL TRIAL: NCT04252209
Title: the Effect of Mixture of Natural Products As Salivary Substitute In Comparison To Carboxy Methyl Cellulose In Treatment Of Xerostomia In Patients With Sjogren's Syndrome: Cross Over Randomized Clinical Trial
Brief Title: the Effect of Mixture of Natural Products As Salivary Substitutes in Treatment Of Xerostomia
Acronym: RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mahmoud abd El kader, Principle investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMD3-7-2 CairoU
Record Dates: First submitted 2020-01-26; First posted 2020-02-05 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Sjogren's Syndrome; Xerostomia
Keywords: xerostomia; oral dryness; dry mouth
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia | interventions — Biological Products

STUDY DESIGN:
Intervention Model Description: 50% of patients will start with intervention (A) for 2 weeks then wash out periods for 7 days then control for 2 weeks and the other 50% will start with control for 2 weeks then wash out periods for 7 days then intervention (B) for 2 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trial participants will be blinded as the two interventions will have the same properties in the same container. The investigator will be blinded as he will not know the treatment assigned for the participants. Also the outcome assessor and the statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with sjogren's received natural mixture (Experimental): The intervention is a moisturizing gel containing 10% aloe vera jelly, 10% coconut oil, 3% peppermint essential oil, 3% carboxy methyl cellulose, 10% propylene glycol, and 0.1% potassium sorbate and water up to 100%.
  applied topically in all surfaces of oral mucosa 4 times daily after eating and before sleep
  Interventions: Other: natural herbs of coconut, aloe vera, and pepperint
- patients with sjogren's recievrd CMC (Active Comparator): the control is a moisturizing gel containing 3% peppermint essential oil, 3% carboxy methyl cellulose, 10% propylene glycol, and 0.1% potassium sorbate and water up to 100%.
  applied topically in all surfaces of oral mucosa 4 times daily after eating and before sleep
  Interventions: Other: carboxy methyl cellulose

INTERVENTIONS:
Other: natural herbs of coconut, aloe vera, and pepperint — mixture of herbal oils of coconut, peppermint, aloe vera
  Other Names: natural products
  Arms: patients with sjogren's received natural mixture
Other: carboxy methyl cellulose — a moisturizing gel contained 3%carboxy methyl cellulose, 3% peppermint essential oil, 10% propylene glycol, 0.1% potassium sorbate, and water up to 100%.
  Other Names: CMC
  Arms: patients with sjogren's recievrd CMC

SUMMARY:
evaluate the efficacy of natural herbal mixture of aloe vera gel, coconut oil and peppermint in comparison to the carboxy methyl cellulose on xerostomia in a sample of patients with Sjogren's syndrome.

DETAILED DESCRIPTION:
The study will be held in the Rheumatology clinic at El Kasr Al-Ainy Cairo University Hospital in patients with Sjogren's syndrome. Population: A random sample of adult patients diagnosed with primary or secondary Sjogren's syndrome attending at the Rheumatology clinic in El Kasr Al-Ainy, Cairo University Hospital will be enrolled in the study in a consecutive order.

The interventions will be in the form of gel to be maintained for long period in the oral cavity. The intervention is a moisturizing gel containing 10% aloe vera jelly, 10% coconut oil, 3% peppermint essential oil, 3% carboxy methyl cellulose, 10% propylene glycol, and 0.1% potassium sorbate and water up to 100%. The control is also a moisturizing gel contained 3%carboxy methyl cellulose, 3% peppermint essential oil, 10% propylene glycol, 0.1% potassium sorbate, and water up to 100%.

Both gels had similar appearance, color, smell, and weight. They will be produced by professional pharmacist in faculty of pharmacy, Al Azher university, Cairo, Egypt.it was taken from previous study with modification in percentage of aloe vera and adding coconut oil. Both gels will be applied topically in all surfaces of oral mucosa 4 times daily after eating and before sleep . The same individuals will deliver the trial interventions in all study groups, both gels will be used for 2 weeks then washout period for 7 days then cross over them. Modification of life style will be promoted as daily tooth brushing, hydration with sufficient amounts of water, eating fibrous food as fruits and vegetables, avoid any alcohol mouth wash or any other topical oral products. The medication will be withdrawn if any allergic reaction occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Patients physically able to participate in the clinical trial.
3. Patients diagnosed with Sjogren's syndrome using 2016 ACR/EULAR classification criteria (Shiboski et al., 2017).
4. Secondary sjogren patients with rheumatoid arthritis.
5. Patients with clinical oral dryness positive scores.

Exclusion Criteria:

1. Patients with previous radiotherapy.
2. Patients not approved to participate in the clinical trial.
3. Patients didn't complain from xerostomia.
4. Patients with diabetes mellitus.
5. Patients taking drugs caused xerostomia as antidepressants, anticholinergics, antihistamines, and anxiolytics and antihypertensives (Campos et al., 2019).
6. Patients with symptomatic oral lesions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
subjective oral dryness | 14 days
  subjective oral dryness measured by bother 1 scale. It is patient centered scale as the patient reported how much he suffer from oral dryness on scale from 1 - 10.as 1 mean mild dryness and 10 mean severe oral dryness

SECONDARY OUTCOMES:
objective oral dryness | 14 days
  using the Challacombe Scale. It will be assessed by the investigator in the first visit (baseline assessments before the interventions) and in the end of two weeks (final assessments).as score 1 mean mild oral dryness and score 10 mean severe oral dryness

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo Univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
efficacy of mixture of aloe vera, coconut and peppermint in treatment of subjective and objective oral dryness
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years

REFERENCES:
- [Result] Atashi V, Yazdannik A, Mahjobipoor H, Ghafari S, Bekhradi R, Yousefi H. The Effects of Aloe vera-Peppermint (Veramin) Moisturizing Gel on Mouth Dryness and Oral Health among Patients Hospitalized in Intensive Care Units: A Triple-Blind Randomized Placebo-Controlled Trial. J Res Pharm Pract. 2018 Apr-Jun;7(2):104-110. doi: 10.4103/jrpp.JRPP_18_21. PMID 30050964